CLINICAL TRIAL: NCT03901885
Title: Impact of Deep Endometriosis Surgery on Sexual Health
Brief Title: Sexual Health After Endometriosis Surgery
Acronym: SSACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0656
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Major women operated for deep endometriosis (Other): Major women operated for deep endometriosis at the Lyon Sud Hospital Center (CHLS) of the Hospices Civils de Lyon (HCL).
  Interventions: Other: Female Sexual Function Index questionnaire

INTERVENTIONS:
Other: Female Sexual Function Index questionnaire — Assessment of FSFI (Female Sexual Function Index) questionnaires preoperatively and postoperatively (4 months).

SUMMARY:
Endometriosis is a disease affecting between 5 and 15% of women and more than 40% of infertile women.

The main stakes of this disease are that it is benign but difficult to diagnose, often very painful, difficult to predict, potentially recurrent, while being resolvable at menopause. It affects women of childbearing age and can cause infertility and pain during intercourse. Also, by its characteristics, it can significantly deteriorate the quality of life.

The management of endometriosis, from diagnosis to treatment, is not consensual. There are medical or surgical treatments depending on the severity of the lesions, their location and the severity of the symptoms. Deep endometriosis, that is to say when there is digestive, urinary, utero sacral or peritoneal ligament more than 5mm deep, poses, in particular, a therapeutic problem because surgery is often the only option but it can be decadent.

Due to genital involvement, this disease has a real impact on the sexuality of patients. Surgery allows in a number of cases to reduce pain, including those occurring during intercourse. But the impact on sexuality in a more global way remains to be studied. The latter can be improved by the reduction of pain, but impacted by the surgery which is not insignificant on the representation of the woman of her own body.

ELIGIBILITY:
Inclusion Criteria:

* Major women operated for deep endometriosis at the Lyon Sud Hospital Center (CHLS) of the Hospices Civils de Lyon (HCL).

Exclusion Criteria:

* Minor patient
* No indication for operation or indication of hysterectomy
* Isolated uterine adenomyosis
* Patient opposing her participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
Consequences of the surgical management of a deep endometriosis on the quality of the sexual life of the patients. | 4 months
  Assessment of FSFI (Female Sexual Function Index) questionnaires preoperatively and postoperatively (4 months).

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Poilblanc, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France